CLINICAL TRIAL: NCT05351281
Title: Appropriate Medication USE in Dutch Terminal Care: AMUSE Trial
Brief Title: Appropriate Medication Use in Dutch Terminal Care
Acronym: AMUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof.dr Carin (C.C.D.) van der Rijt (Other)
Collaborators: Rijnstate Hospital (Other); Ikazia Hospital, Rotterdam (Other); Noordwest Ziekenhuisgroep (Other); Laurens Cadenza Zuid (Unknown); Nijmegen University Academic Network Family Medicine (Network); Gezondheidscentrum Krimpen (Unknown)
Responsible Party: Sponsor-Investigator, Prof.dr Carin (C.C.D.) van der Rijt, Professor Palliative Oncology of Department Medical Oncology, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NL7830507821; MEC-2021-0624 (Other: Ethics Committee)
Record Dates: First submitted 2022-04-11; First posted 2022-04-28 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Palliative Care; Terminal Care; Medication Therapy Management; Clinical Decision Support System (CDSS); Quality of Life

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized study. The stepped-wedge design involves random and sequential crossover of 7 clusters (=7 different study sites) from the control to the intervention group, until all clusters are exposed. All clusters will start as control sites, where care is provided as usual. Every twelve weeks, one site will crossover from control to intervention group
Masking Description: Sites will crossover from control to the intervention group in a random order. During the study all parties have knowledge of the interventions assigned to individual participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients in the standard of care arm will receive the usual treatment
- CDSS-OPTIMED (Experimental): In the experimental arm, attending physicians will receive weekly medication alerts from the Clinical Decision Support System (CDSS) within 1 week after inclusion of the patient. The CDSS-OPTIMED will send a medication advice on a weekly basis, based on a weekly analysis of patient's medication. The medication alerts will be sent to the physician's email address. The physician is free to follow or ignore the advice in the alerts. If the physicians thinks these alerts are relevant for the patient, the physician will discuss these alerts with the patient and/or relatives. After this conversation, the physician will prescribe or deprescribe medications based on the alerts.
  Interventions: Device: CDSS-OPTIMED

INTERVENTIONS:
Device: CDSS-OPTIMED — The CDSS-OPTIMED is a software program that provides the physician with a personalized alert on whether to consider stopping or starting medication for a specific patient with a life expectancy of less than 3 months.
  Arms: CDSS-OPTIMED

SUMMARY:
The AMUSE trial is a multicentre stepped-wedge cluster randomized controlled trial where medication optimization of patients with a life expectancy of less than three months is investigated by using CDSS-OPTIMED (a personalized medication advice to attending physicians of patients in the last phase of life) The investigators will include 250 patients, in 7 different study sites across the Netherlands. The primary outcome is an assessment of the quality of life of patients, two weeks after baseline assessment.

DETAILED DESCRIPTION:
Rationale: patients in the last phase of life often use many medications that are continued until shortly before they die. This is partly inevitable, because these patients often experience multiple distressing symptoms. However, for a considerable number of medications currently often used at the end of life, the benefit is debatable, e.g. because they are aimed at the long-term prevention of illness.

Primary objective: to examine whether the use of CDSS-OPTIMED, a personalized medication advice to attending physicians of patients in the last phase of life, contributes to patients' quality of life.

Main study endpoints: the primary endpoint is patients' quality of life two weeks after baseline assessment, as measured by the EORTC QLQ-C15-PAL questionnaire (scale 0 to 100).

Potential risks and benefits associated with participation: the intervention in this trial supports physicians in using available evidence and knowledge when deprescribing medication for patients in the last phase of life. The intervention does not involve experimental treatment or medication. The investigators expect no other risks than known side effects of (stopping) medications. The investigators are aware that the trial population concerns vulnerable people who may experience fluctuating symptoms and levels of suffering across their disease trajectory. The investigators acknowledge the risk of overburdening participants. If patients feel burdened by participating in the study, they are encouraged to indicate that.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older and provides informed consent to participate.
* The patient is aware that recovering from his/her disease is unlikely, to be assessed by the attending physician.
* The patient is competent to decide about trial participation
* The patient has a life expectancy of at least two weeks and at most three months, as estimated by an attending physician.

Exclusion Criteria:

* The patient is incapable of filling in a questionnaire (patients may be supported by relatives when filling in the questionnaire).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Patients' quality of life | Two weeks after baseline assessment
  Measured by the quality of life question of the European Organization for Research and Treatment of Cancer Quality of Life Group 15 item core questionnaire for palliative care ( = EORTC QLQ-C15-PAL questionnaire)
  Scale 1 to 7. Scale minimum 1 (very poor). Scale maximum 7 (excellent).
  Score will be rescaled to a scale from 0 to 100, in which 100 is an excellent outcome

SECONDARY OUTCOMES:
Patients' quality of life | At day 7, 21, 28, and then every 28 days until death, with a maximum of 24 weeks,
  Measured by the quality of life question of the European Organization for Research and Treatment of Cancer Quality of Life Group 15 item core questionnaire for palliative care ( = EORTC QLQ-C15-PAL questionnaire)
  Scale 1 to 7. Scale minimum 1 (very poor). Scale maximum 7 (excellent).
  Score will be rescaled to a scale from 0 to 100, in which 100 is an excellent outcome
Symptoms and the occurrence of potential side effects of continuing or discontinuing medication | At day 1-7, 14, 21, 28, and then every 28 days until death, with a maximum of 24 weeks
  Assessed by the Utrecht Symptoom Dagboek (USD, which is based on the Edmonton Symptom Assessment Scale (ESAS))
  Scale 0 to 10. Scale minimum 0 (no symptoms). Scale maximum 10 (worst possible symptoms)
Systolic and Diastolic Blood Pressure (mmHg) in case of using antihypertensives (continued or discontinued) | At day 1-7, 14, 21, 28, and then every 28 days until death, with a maximum of 24 weeks
  Measured by patients' attending health care professional
Glucose level (mmol/L) in case of using antidiabetics (continued or discontinued) | At day 1-7, 14, 21, 28, and then every 28 days until death, with a maximum of 24 weeks
  Measured by patients' attending health care professional
Occurence of thrombo-embolic and bleeding events | From inclusion until death, with a maximum of 24 weeks
  Measured and reported in the data management system by the time between inclusion and death
Time spent on discussing the medication with the patient | From inclusion until death, with a maximum of 24 weeks
  As registered in the electronic patient files on a time scale (0-5 minutes, 6-10 minutes, 11-15 minutes, 16-20 minutes, >21minutes) Scale minimum: 0-5 minutes (short). Scale maximum: >21 minutes (long)
Health care costs | Retrospectively over full study period (From inclusion until death, with a maximum of 24 weeks)
  Measured by using a medical file checklist. Items to be assessed include: medication prescriptions, hospital admissions and in-hospital care
Medication prescriptions (All medication used by the patient during te whole study period) | From inclusion until death, with a maximum of 24 weeks
  Measured by using a medical file checklist in our data management system. Derived from patients' medical records and the pharmacist's information system
Patient survival | From inclusion until death, with a maximum of 24 weeks
  Derived from patients' medical records and contact with the patient

OTHER OUTCOMES:
Costs of the intervention | Retrospectively over full study period. Full study period is from inclusion until death, with a maximum of 24 weeks.
  Development and training costs (proformas completed by the developers and the study personnel).
  Operational costs (including time spent on discussing medication alerts with the pharmacist and patient/relative derived from patients' medical records. And time registrations via automated system extracts, derived from CDSS-OPTIMED)

CONTACTS AND LOCATIONS:
Overall Officials: Carin van der Rijt, Prof, MD, Principal Investigator — Erasmus Medical Center; Eric Geijteman, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (7):
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Rijnstate Hospital, Arnhem
  - Gezondheidscentrum Krimpen, Krimpen aan den IJssel
  - Nijmegen University Academic Network Family Medicine, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Laurens Cadenza Zuid, Rotterdam

IPD SHARING:
Plan to Share IPD: No
Individual participant data will already be shared with the Dutch national centre of expertise and repository for research data (DANS)

REFERENCES:
- [Derived] van Hylckama Vlieg MAM, Pot IE, Visser HPJ, Jong MAC, van der Vorst MJDL, van Mastrigt BJ, Kiers JNA, van den Homberg PPPH, Thijs-Visser MF, Oomen-de Hoop E, van der Heide A, van der Kuy PHM, van der Rijt CCD, Geijteman ECT. Appropriate medication use in Dutch terminal care: study protocol of a multicentre stepped-wedge cluster randomized controlled trial (the AMUSE study). BMC Palliat Care. 2024 Jan 3;23(1):6. doi: 10.1186/s12904-023-01334-x. PMID 38172930